CLINICAL TRIAL: NCT01184404
Title: Bosentan Improves Clinical Outcome of Adults With Congenital Heart Disease or Mitral Valve Lesions Who Undergo CArdiac Surgery
Acronym: BOCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Berto J Bouma (Other)
Responsible Party: Sponsor-Investigator, Berto J Bouma, MD PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03603
Record Dates: First submitted 2010-08-11; First posted 2010-08-19 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Congenital Heart Disease
Keywords: Congenital heart disease; Cardiac surgery; Bosentan
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Bosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): The treatment group receives a starting dose of 62.5 mg tablet bosentan twice daily for four weeks followed by 125 mg tablet of bosentan twice daily two weeks prior to and 12 weeks after surgery.
  Interventions: Drug: Bosentan
- Control (No Intervention)

INTERVENTIONS:
Drug: Bosentan — The treatment group receives a starting dose of 62.5 mg tablet bosentan twice daily for four weeks followed by 125 mg tablet of bosentan twice daily two weeks prior to and 12 weeks after surgery.
  Other Names: Tracleer Bosentan
  Arms: Treatment

SUMMARY:
Cardiac surgery relieves symptoms and increases life expectancy in cardiac patients, with and without congenital heart disease (CHD). However, cardiac surgery involves many risks of complications, such as bleeding, arrhythmias, and death.Right ventricular failure is another complication, contributing to poor clinical outcome. Right ventricular failure is a clinical syndrome, often difficult to treat, characterized by edema, elevated jugular venous pressure, oliguria, hypotension, and in severe cases shock, multi organ failure and death. Patients with CHD and patients with mitral valve lesions are suspected to be at increased risk for developing right ventricular failure post-operatively. In addition, other clinical factors contributing to right ventricular failure are mechanical pulmonary ventilation, pulmonary hypertension and cardiac surgery. Right ventricular failure during cardiac surgery is caused by the cardiopulmonary bypass by reperfusion with high partial pressures of oxygen, air embolism, and the release of cytokines. The endothelin-1 cytokine induces vasoconstriction of the pulmonary arterioles resulting in right ventricular afterload elevation. Treating patients with an endothelin-1 receptor antagonist might improve clinical outcome post operatively by decreasing right ventricular afterload

DETAILED DESCRIPTION:
Rationale: Cardiac surgery relieves symptoms and increases life expectancy in cardiac patients, with and without congenital heart disease (CHD). However, cardiac surgery involves many risks of complications, such as bleeding, arrhythmias, and death. Right ventricular failure is another complication, contributing to poor clinical outcome. This clinical syndrome is often difficult to treat and is characterized by edema, elevated jugular venous pressure, oliguria, hypotension, and in severe cases shock, multi organ failure and death.

Patients at increased risk for developing post operative right ventricular failure are those with CHD or with mitral valve lesions, because of their elevated afterload. Other clinical factors contributing to right ventricular failure are mechanical pulmonary ventilation, pre-existing pulmonary hypertension and cardiac surgery. Right ventricular failure due to cardiac surgery is caused by the cardiopulmonary bypass, by reperfusion with high partial pressures of oxygen, air embolism, and the release of cytokines. The endothelin-1 cytokine release during cardiac surgery induces vasoconstriction of the pulmonary arterioles resulting in right ventricular afterload elevation. Therefore, we hypothesize that treating patients with an endothelin-1 receptor antagonist will improve clinical outcome, measured by aerobic capacity (peak V'O2), by decreasing right ventricular afterload peri-operatively.

Objective: To investigate whether an endothelin-1 receptor antagonist improves aerobic capacity (peak V'O2) in adults with CHD or with mitral valve lesions who undergo cardiac surgery.

Study design: A prospective randomized open label assessment with blinded end-points (PROBE-design). Total duration of the study is 18 weeks with 6 weeks pre-operative and 12 weeks post-operative treatment with bosentan.

Study population: Adults with CHD who undergo cardiac surgery and patients undergoing mitral valve surgery in the Academic Medical Centre in Amsterdam. Patients will be randomized six weeks before surgery. The study will continue until 12 weeks postoperatively.

Intervention: The treatment group receives a starting dose of 62.5 mg tablet bosentan twice daily for four weeks followed by 125 mg tablet of bosentan twice daily two weeks prior to and 12 weeks after surgery. The other group receives no study medication.

Main study parameters/endpoints: 1) on the intensive care unit a) hemodynamics b)Sequential Organ Failure Assessment (SOFA) score and c) hours of hospitalization 2) at discharge the right ventricular function (assessed by transthoracic echocardiography) 3) six weeks post-operatively a) clinical condition with exercise capacity (peak V'O2) b) right ventricular function (assessed by transthoracic echocardiography) c) the quality of life 4) twelve weeks post-operatively a) right ventricular function (assessed by transthoracic echocardiography) b) differences in clinical status and symptoms

ELIGIBILITY:
Inclusion Criteria:

* Adults with CHD or mitral valve lesions who are scheduled for elective cardiac surgery

Exclusion Criteria:

* Current treatment with bosentan
* Systemic arterial pressure < 85 mmHg
* Incapable of giving informed consent
* Hypersensitivity to bosentan or any of its help substances
* Moderate to severe liver disease: Child-Pugh class B or C
* Raised plasma transaminases level > three times limiting value.
* Simultaneous use of cyclosporine A
* Percutaneous Transluminal Angioplasty procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-09; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
peak V'O2 | 18 weeks
  The primary objective of this study is to determine changes in aerobic capacity (peak V'O2)in adult CHD patients or with mitral valve lesions who undergo surgery comparing treated with non-treated patients.

SECONDARY OUTCOMES:
Right ventricular function | 18 weeks
  To determine 18 weeks after baseline differences in right ventricular function (assessed by transthoracic echocardiography)

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands